CLINICAL TRIAL: NCT00119704
Title: Treatment of Lateral Epicondylitis With Botulinum Toxin: A Randomized Controlled Trial
Brief Title: Treatment of Tennis Elbow With Botulinum Toxin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: New World Development Company Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2002.354-T
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2006-05-09 (Estimated); Status verified 2005-06

CONDITIONS: Epicondylitis, Lateral Humeral
MeSH Terms: conditions — Tennis Elbow | interventions — Botulinum Toxins, Type A; Saline Solution

INTERVENTIONS:
Drug: Botulinum toxin A injection or normal saline

SUMMARY:
The purpose of this study is to determine whether Botulinum A toxin is effective in the treatment of tennis elbow (lateral epicondylitis).

DETAILED DESCRIPTION:
Tennis elbow (lateral epicondylitis) is a common cause of chronic elbow pain and wrist extensor dysfunction in adults, affecting 1% to 3% of the general population per year.

There is currently no consensus on its optimal treatment with wide-ranging options available. The best available scientific evidence suggests that only topical non-steroidal anti-inflammatory drugs and possibly, oral non-steroidal anti-inflammatory drugs may be useful for short term pain relief, while corticosteroid injections presented both benefits and harms as a short term measure.

Botulinum toxin has been reported in the treatment of lateral epicondylitis with promising results but these studies lack a control group bringing up the question whether recovery was a result of intervention or the natural history of the disease.

Method:

A twin-center, prospective, randomized, double-blind, placebo-controlled trial in which all patients received either a botulinum injection or a placebo saline injection.

Consecutive patients over 18 years old with tennis elbow referred to the outpatient clinic at the investigators' institution will be screened for this study. Eligible patients will be invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and up
* Pain at the lateral side of the elbow
* Pain at the lateral epicondyle during resisted dorsiflexion of the wrist with the elbow in full extension
* Pain for longer than 3 months

Exclusion Criteria:

* Previous operations (including previous steroid injections for the disorder)
* Nerve entrapment
* Pregnancy and while breast-feeding
* Presence of systemic neuromuscular disorders such as myasthenia gravis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-09; Study Completion 2005-03

PRIMARY OUTCOMES:
100 mm visual analog scale (VAS)

SECONDARY OUTCOMES:
Grip strength measured with a Jamar Hydraulic Hand Dynamometer with the elbow fully extended and the hand in middle position.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew CF Hui, MRCP, Principal Investigator — Department of Medicine & Therapeutics, Facutly of Medicine, The Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, New Territories
  - North District Hospital, Sheung Shui, New Territories

REFERENCES:
- [Result] Wong SM, Hui AC, Tong PY, Poon DW, Yu E, Wong LK. Treatment of lateral epicondylitis with botulinum toxin: a randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2005 Dec 6;143(11):793-7. doi: 10.7326/0003-4819-143-11-200512060-00007. PMID 16330790